CLINICAL TRIAL: NCT04092998
Title: Histopathological Changes and Surgical Complications in Thermocautery Circumcision
Brief Title: Circumcision With Use of Thermocautery and Histopathological Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed gamal, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Circumcision
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Circumcision

STUDY DESIGN:
Intervention Model Description: male infant presented for Circumcision
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermocautery VS scalpel circumcision (Experimental): Thermocautery circumcision in comparison to circumcision with traditional scalpel
  Interventions: Procedure: Thermocautery circumcision

INTERVENTIONS:
Procedure: Thermocautery circumcision — Histopathological changes from thermocautery circumcision
  Other Names: scalpel circumcision

SUMMARY:
Histo pathological changes that occurs in thermo cautery circumcision and the range of damage prepuce from thermal effect in comparison with scalpel circumcision

DETAILED DESCRIPTION:
Circumcision is one of the most commonly performed surgical procedures worldwide. It is known that more than one million children are circumcised annually in the USA alone . Moreover, the WHO has begun to recommend circumcision on the basis of studies indicating its positive effects on human health and especially its role in protection from AIDS . Because of this, thousands of people have been circumcised by many migratory circumcision teams, especially in Africa.

Considering that 1 200 000 children are born annually in Turkey and 51% of them are male, on the basis of data from the Turkish Institute of Statistics, it may be speculated that about 60 000 circumcisions are performed annually in Turkey.

However, the circumcision procedure cannot be performed in health institutions as a routine procedure because of health regulations. When the Social Security Institute incorporated circumcision into the social insurance coverage in 2007, it led to circumcision being performed in the health institutions. Health institutions that were already burdened cannot meet the demands for circumcision. Thus, the search has begun for faster and reliable circumcision techniques with fewer complications. The present study aimed to compare bipolar thermal cautery-assisted circumcision technique, considered to be capable of meeting such demands, with the classical circumcision technique.

Aim of Work This study is aiming to assess the outcome of using thermo cautery in circumcision

Surgical Steps:

small skin incision over prepuce by thermo cautery

stitching if there is bleeding

Insertion of a urinary catheter if suspect uretheral injury

ELIGIBILITY:
Inclusion Criteria:

* all male gender

Exclusion Criteria:

* females
* micro penis
* hypospedias
* epispedias
* ambigilious genitalia

Min Age: 40 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male infant
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
early wound complications | 1 week
  wound infection (with or without removal of the mesh) wound necrosis wound hematoma bleeding
late wound complications | 1 month
  wound infection (with or without removal of the mesh) wound necrosis wound hematoma

CONTACTS AND LOCATIONS:
Overall Officials: gamal makhlouf, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age , sex , clinical diagnosis
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: age , sex , clinical diagnosis